CLINICAL TRIAL: NCT00820716
Title: Comparison of Two Types of Exercise Training for Asthmatic Subjects : Interests and Limits
Brief Title: Exercise Training in Asthma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in recruiting patient
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3825; 2006-A00090-51
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2011-08

CONDITIONS: Asthma
Keywords: Asthma; Asthmatic subjects; Exercise training; Constant load; Alternate load
MeSH Terms: conditions — Asthma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CA (Experimental): Exercise training with alternate load
  Interventions: Other: Exercise training
- CC (Active Comparator): Exercise training with constant load
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — Comparison of two methods of exercise training: alternate load versus constant load realized at moderate or high intensities

SUMMARY:
The aim of the study is to compare two methods of exercise training: alternate load versus constant load realized at moderate or high intensities, in order to define the interests and the limits of each one of these two methods. The finality is to make possible to the expert to choose what exercise training induces the best results quickly and to make its choice according to the therapeutic objectives which it lays down.We also evaluate the effects of these exercises training on the vagal response and the bronchial tone of the asthmatics. From a clinical point of view, a close attention will be paid to the effects of these exercises training on the control of asthma and the quality of life of the subjects

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old
* mild to moderate persistent asthma (GINA classification)
* stabilized asthma
* physical activity level between 5 and 11 (Baecke and coll, 1982)
* no contra-indication for physical training

Exclusion Criteria:

* cardiovascular pathology
* metabolic pathology
* traumatic pathology
* BMI≥30
* tobacco
* diabetes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2009-09-21 (Actual); Primary Completion 2010-10-15 (Actual); Study Completion 2010-10-15 (Actual)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2max) | At T-1 = eight weeks before training - At T0 = beginning of training - At T1 = eight weeks after training
Maximal power output (Pmax) | At T-1 = eight weeks before training - At T0 = beginning of training - At T1 = eight weeks after training

SECONDARY OUTCOMES:
Exhaled NO (eNO) | At T-1 = eight weeks before training - At T0 = beginning of training - At T1 = eight weeks after training
Heart rate variability | At T-1 = eight weeks before training - At T0 = beginning of training - At T1 = eight weeks after training
Force Expiratory Volume in one second (FEV1) | At T-1 = eight weeks before training - At T0 = beginning of training - At T1 = eight weeks after training

CONTACTS AND LOCATIONS:
Overall Officials: Evelyne LONSDORFER, MD, Study Director — Hôpitaux Universitaires de Strasbourg
Locations (2):
- France (2):
  - Service de Physiologie et d'Explorations Fonctionnelles - Pôle de Pathologie Thoracique - Nouvel Hôpital Civil, Strasbourg
  - Service de Pneumologie - Pôle de Pathologie Thoracique - Nouvel Hôpital Civil, Strasbourg